CLINICAL TRIAL: NCT03041220
Title: Best Incision Site for Obese Patients - Low Versus High Transverse
Status: Withdrawn | Type: Observational
Why Stopped: PI no longer at institution
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 24387
Record Dates: First submitted 2017-01-11; First posted 2017-02-02 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cesarean section: Obese pregnant patients who have had a cesarean section.
  Interventions: Procedure: cesarean section

INTERVENTIONS:
Procedure: cesarean section — obese patients (BMI of 30 or greater) who have had a cesarean section

SUMMARY:
Retrospective chart review using both out patient and inpatient records of obese patients (BMI of 30 or greater) who have had a cesarean section since the year 2009. We will evaluate the patient's BMI, their skin incision type at time of c-section, their co-morbidities, number of previous c-sections and post partum follow up for wound infection, wound separation and wound breakdown. We will also review operative notes to evaluate blood loss, length of surgery and complications during surgery. We will obtain maternal characteristics and information about the pregnancy.

DETAILED DESCRIPTION:
Past studies have looked primarily at vertical vs low transverse skin incision. There is data that performing a high transverse skin incision on obese patients leads to better visualization and less wound infection but there are few studies comparing it directly to low transverse skin incision.

Retrospective chart review of obese patient's who have had a cesarean section at St Mary's hospital by either a low or high transverse skin incision between January 1, 2009 - July 31, 2014. We will review charts up to 6 week postpartum.

Pregnancies will be identified through identifing those who have cesarean sections. They will be narrowed down by those who have BMI of > 30. Maternal prenatal records, postnatal records and delivery records will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* obese patients (BMI of 30 or greater) who have had a cesarean section

Exclusion Criteria:

* Vaginal delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ages between 18 - 45 years, female, and no limitation on ethnic background.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Type of skin incision | Delivery to 6 weeks postpartum
  Identify which type of skin incision has better outcomes in obese pregnant patients

CONTACTS AND LOCATIONS:
Overall Officials: Heather Said, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No